CLINICAL TRIAL: NCT01971346
Title: The Immunological Basis for Treatment Resistance to Anti-TNF Treatments
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Johann E Gudjonsson MD, PhD, Assistant Professor of Dermatology, Medical School, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Derm 652
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Results first posted 2019-01-09 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Psoriasis
Keywords: Psoriasis; ENBREL; etanercept; anti-TNF
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etanercept (Other): 100 mg Etanercept injections per week for 3 months.
  Interventions: Drug: etanercept

INTERVENTIONS:
Drug: etanercept — 100 mg Etanercept injections per week (2 separate single-use pre-filled 50 mg subcutaneous injections taken on two separate days) for 3 months
  Other Names: ENBREL

SUMMARY:
The purpose of this study is to determine the relationship between two types of cell signals, type I interferon (IFN) and tumor necrosis factor (TNF), in psoriatic skin prior to and during treatment with etanercept and correlate that information with the degree of the improvement in the psoriasis.

DETAILED DESCRIPTION:
Hypothesis: The balance between type I IFN and TNF determines the response to anti-TNF treatment. The goal of the proposed study is to address this hypothesis and demonstrate that the strength of the type I IFN signature in psoriatic skin is the major determinant of the clinical response to anti-TNF treatment.

Purpose: Determine the strength of the type I interferon and TNF signal in psoriatic skin prior to and during treatment with etanercept and correlate with degree of clinical improvement.

Study Population: up to 50 subjects, men or women over the age of 18 with clinically stable plaque psoriasis, who meet the wash out requirements and other exclusion criteria

Psoriatic patients will receive 100 mg etanercept per week (2 separate single-use pre-filled 50 mg subcutaneous injections taken on two separate days) for 3 months.

Procedures: Urine pregnancy test, TB test, photography, Physical Examinations, Skin Examinations, Study Drug, Peripheral blood and biopsies

Anticipated Results: We expect that patients with strong IFN-α signature in psoriatic skin along with weak TNF-α signature will have minimal response to anti-TNF treatment, while patients with the opposite pattern, weak IFN and strong TNF signature, will have significant clinical improvement.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at screening.
* Clinically stable moderate to severe plaque psoriasis at screening and baseline.
* Subject must be:

  * A man or
  * A woman who is surgically sterile or at least 3 years postmenopausal or
  * A woman of childbearing potential who has had a negative pregnancy test within 7 days before the first dose of study drug.
* If the subject is sexually active, (s)he must agree to use a medically acceptable form of contraception during screening and throughout the study.

Exclusion Criteria:

* Grade 3 or 4 adverse events or infections within 28 days before screening, or between the screening visit and drug initiation.
* Active or chronic infection within 4 weeks before screening visit, or between the screening and baseline visits.
* Evidence of skin conditions other than psoriasis that would interfere with the evaluations of the effect of study medication on psoriasis.
* Use of oral psoralen with ultraviolet A (PUVA), oral retinoids, cyclosporine, alefacept, or any other systemic anti-psoriasis therapy within 28 days study drug initiation.
* Use of ulltraviolet B (UVB) therapy, topical steroids at no higher than moderate strength, topical vitamin A or D analog preparations, or anthralin with 14 days of study initiation.
* Prior or concurrent use of cyclophosphamide therapy
* Concurrent sulfasalazine therapy.
* Known hypersensitivity to Enbrel® (etanercept) or any of its components or known to have antibodies to etanercept.
* Current enrollment in any other investigational device or investigational drug trial(s), or receipt of any other investigational agent(s) within 28 days before baseline visit.
* Use of any biologic drugs within 28 days of study drug initiation.
* Concurrent use of Anakinra.
* Severe comorbidities (diabetes mellitus requiring insulin; congestive heart failure (CHF) of any severity or myocardial infarction or cerebrovascular accident or transient ischemic attack within 3 months of screening visit; unstable angina pectoris, uncontrolled hypertension (sitting systolic blood pressure (BP) <80 mm Hg or > 160 or diastolic BP > 100 mm Hg), oxygen-dependent severe pulmonary disease, history of cancer within 5 years (other than resected cutaneous basal or squamous cell carcinoma of the skin or in situ cervical cancer)
* Known history of tuberculosis (TB), or previous positive purified protein derivative (PPD) test. Any mycobacterial disease or high risk factors for tuberculosis (TB), such as family member with TB, positive purified protein derivative (PPD) or taking anti-tuberculosis medication.
* Known HIV-positive status or known history of any other immuno-suppressing disease.
* Concurrent or history of psychiatric disease that would interfere with ability to comply with study protocol or give informed consent.
* History of alcohol or drug abuse within 12 months of screening visit.
* Latex sensitivity [Nota Bene: only applicable if they are using prefilled syringe or prefilled SureClick™ autoinjector presentations]
* Exposure to hepatitis B or hepatitis C or to high risk factors for hepatitis B or C, such as intravenous drug use in patient.
* Systemic lupus erythematosus, history of multiple sclerosis, transverse myelitis, optic neuritis or seizure disorder.
* Use of a live vaccine 90 days prior to screening visit, or concurrent use of a live vaccine.
* Any condition or circumstances judged by the patient's physician[or the investigator or medically qualified study staff] to render this clinical trial detrimental or otherwise unsuitable for the patient's participation.
* History of non-compliance with other therapies.
* Pregnant or nursing females.
* Diagnosis of multiple sclerosis in first degree family relationship (parent, sibling or child)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03-13 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johann Gudjonsson, MD PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Department of Dermatology, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Etanercept
Started | 50 (Four subjects signed the informed consent and terminated the study before beginning.)
Completed | 42
Not Completed | 8
Not completed — Protocol Violation | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Of the 50 subjects enrolled, four subjects terminated the study after signing the informed consent, yet before beginning the study.
Arm/Group | Etanercept
Number analyzed (Participants) | 46
Age, Continuous [Mean (Full Range); unit: years] | 40.83 [19 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 44
  More than one race | 1
  Unknown or Not Reported | 0
Psoriasis Area and Severity Index (PASI) Score [Mean (Full Range); unit: units on a scale] — The Psoriasis Area and Severity Index is the industry standard to decrease/eliminate subjectivity in determining psoriasis severity. It is a quantitative rating scale for measuring the severity of psoriatic lesions based on area coverage and plaque appearance. The severity of plaque characteristics (erythema, thickness and scaling) for body regions (head, upper limbs, trunk and lower limbs) is combined with the degree of plaque involvement in each body region to determine a single PASI score in the range of 0 (no disease) and 72 (maximal disease).
  units on a scale | 14.16 [3.6 to 42]
Tumor Necrosis Factor (TNF)-alpha Signal [Mean (Full Range); unit: rpkm] — The specified units are the gene expression units and represents Reads per kilobase of region per million mapped reads (RPKM). Population: Biopsy not completed on one subject. Tissue was not worked up/unable to be processed for two subjects.
  rpkm
    number analyzed (Participants) | 43
    (all) | 111.33 [50.45 to 219.31]
Interferon (IFN)-alpha Signal [Mean (Full Range); unit: rpkm] — The specified units are the gene expression units and represents Reads per kilobase of region per million mapped reads (RPKM). Population: Biopsy not completed on one subject. Tissue was not worked up/unable to be processed for two subjects.
  rpkm
    number analyzed (Participants) | 43
    (all) | 2118.20 [1677.65 to 2600.50]

OUTCOME MEASURES:

1. Primary Outcome: Change in Psoriasis Area and Severity Index (PASI) Score
Description: A cumulative change in PASI score from baseline to week 12 will be calculated for each patient. The PASI is the industry standard to decrease/eliminate subjectivity in determining psoriasis severity. It is a quantitative rating scale for measuring the severity of psoriatic lesions based on area coverage and plaque appearance. The severity of plaque characteristics (erythema, thickness and scaling) for body regions (head, upper limbs, trunk and lower limbs) is combined with the degree of plaque involvement in each body region to determine a single PASI score in the range of 0 (no disease) and 72 (maximal disease).
Time Frame: Baseline, 12 weeks
Population: Only those subjects who finished the study (have a Week 0 and Week 12 visit with recorded PASI) are included in the analysis assessing a change from baseline.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- PASI Score at Week 0: PASI will be measured at the baseline visit before treatment.
- PASI Score at Week 12: PASI will be measured at the Week 12 visit after the course of etanercept treatment.
Arm/Group | PASI Score at Week 0 | PASI Score at Week 12
Number analyzed (Participants) | 42 | 42
units on a scale | 13.92 (1.11) | 4.43 (0.48)
Statistical Analysis 1: Comparison: PASI Score at Week 0 vs PASI Score at Week 12; A cumulative score reflecting change in PASI during the course of treatment was calculated and treated as a continuous response variable. Linear modeling was done to determine if change in PASI score was associated with the baseline TNF-alpha signal, baseline IFN-alpha signal and/or an interaction between these two signals; Test type: Other; p = 0.38, Regression, Linear — Type III TNF-alpha p-value=0.36. Type III IFN-alpha p-value=0.36. Interaction was not included in this model

2. Secondary Outcome: Tumor Necrosis Factor (TNF)-Alpha Signal Strength
Description: Strength of TNF-alpha signatures will be measured in skin of study subjects at initiation, during and after treatment. The strength of these signals will be done using bioinformatic approach quantifying transcriptional signature of these cytokines. The strength of the cytokine signals will be treated as a response variable in a univariate repeated measure analysis of variance, with PASI response profile and time as covariates. PASI response profile will be categorized according to improvement in PASI score: responders (greater than 75% reduction in PASI from baseline), intermediate-responders (those with greater than 25% and less than 75% reduction in PASI from baseline), and non-responders (less than 25% reduction in PASI from baseline).
Time Frame: Baseline, Week 6, Week 12
Population: PASI response profile is only done for those subjects who completed the study, n=42. Biopsy not completed on one subject at baseline. Tissue not able to be processed for two subjects at baseline, Week 6 and Week 12. Biopsy not completed on three subjects at Week 6 visit. Biopsy not completed on three different subjects at Week 12 visit.
Measure: Least Squares Mean (Standard Error); unit: rpkm
Groups:
- TNF-alpha Signal Strength at Week 0: Strength of TNF-alpha signature measured in skin of study subjects at Week 0.
- TNF-alpha Signal Strength at Week 6: Strength of TNF-alpha signature measured in skin of study subjects at Week 6.
- TNF-alpha Signal Strength at Week 12: Strength of TNF-alpha signature measured in skin of study subjects at Week 12.
Arm/Group | TNF-alpha Signal Strength at Week 0 | TNF-alpha Signal Strength at Week 6 | TNF-alpha Signal Strength at Week 12
Number analyzed (Participants) | 39 | 37 | 37
rpkm
  PASI Responder: number analyzed (Participants) | 16 | 15 | 15
  PASI Responder | 98.26 (7.40) | 85.82 (10.34) | 64.157 (8.99)
  PASI Intermediate-Responder: number analyzed (Participants) | 20 | 19 | 19
  PASI Intermediate-Responder | 107.79 (6.04) | 108.02 (8.44) | 92.01 (7.34)
  PASI Non-Responder: number analyzed (Participants) | 3 | 3 | 3
  PASI Non-Responder | 110.62 (14.79) | 103.68 (20.67) | 123.08 (17.98)
Statistical Analysis 1: Comparison: TNF-alpha Signal Strength at Week 0 vs TNF-alpha Signal Strength at Week 6 vs TNF-alpha Signal Strength at Week 12; The strength of the TNF-alpha cytokine signals will be treated as a response variable in a univariate repeated measure analysis of variance, with PASI response profile and time as covariates. Testing if TNF-alpha signals are significantly altered during the course of etanercept therapy and if such changes differ between subjects with different PASI response profiles; Test type: Other; p = 0.03, ANOVA — Test of Hypotheses for Between subject effect of PASI profile p-value=0.03 Test of Hypotheses for Within subject effect of Time p-value=0.38 Test of Hypotheses for Within subject effect of Time*PASI profile p-value=0.31

3. Secondary Outcome: Interferon (IFN)-Alpha Signal Strength
Description: Strength of IFN-alpha signatures will be measured in skin of study subjects at initiation, during and after treatment. The strength of these signals in skin will be done using bioinformatic approach quantifying transcriptional signature of these cytokines. The strength of the cytokine signals will be treated as a response variable in a univariate repeated measure analysis of variance, with PASI response profile and time as covariates. PASI response profile will be categorized according to improvement in PASI score: responders (greater than 75% reduction in PASI from baseline), intermediate-responders (those with greater than 25% and less than 75% reduction in PASI from baseline), and non-responders (less than 25% reduction in PASI from baseline).
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: rpkm
Groups:
- IFN-alpha Signal Strength at Week 0: Strength of IFN-alpha signature measured in blood and skin of study subjects at Week 0.
- IFN-alpha Signal Strength at Week 6: Strength of IFN-alpha signature measured in blood and skin of study subjects at Week 6.
- IFN-alpha Signal Strength at Week 12: Strength of IFN-alpha signature measured in blood and skin of study subjects at Week 12.
Arm/Group | IFN-alpha Signal Strength at Week 0 | IFN-alpha Signal Strength at Week 6 | IFN-alpha Signal Strength at Week 12
Number analyzed (Participants) | 39 | 37 | 37
rpkm
  PASI Responder: number analyzed (Participants) | 16 | 15 | 15
  PASI Responder | 2082.72 (70.73) | 2146.83 (84.18) | 2180.36 (88.46)
  PASI Intermediate-Responder: number analyzed (Participants) | 20 | 19 | 19
  PASI Intermediate-Responder | 2106.72 (57.75) | 2186.17 (68.73) | 2107.22 (72.23)
  PASI Non-Responder: number analyzed (Participants) | 3 | 3 | 3
  PASI Non-Responder | 2102.64 (141.46) | 2035.94 (168.36) | 1923.33 (176.92)
Statistical Analysis 1: Comparison: IFN-alpha Signal Strength at Week 0 vs IFN-alpha Signal Strength at Week 6 vs IFN-alpha Signal Strength at Week 12; The strength of the IFN-alpha cytokine signals will be treated as a response variable in a univariate repeated measure analysis of variance, with PASI response profile and time as covariates. Testing if IFN-alpha signals are significantly altered during the course of etanercept therapy and if such changes differ between subjects with different PASI response profiles; Test type: Other; p = 0.34, ANOVA — Test of Hypotheses for Between subject effect of PASI profile p-value=0.34 Test of Hypotheses for Within subject effect of Time p-value=0.73 Test of Hypotheses for Within subject effect of Time*PASI profile p-value=0.57

4. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Response Profile
Description: Subjects will be categorized according to improvement in Psoriasis Area and Severity Index (PASI) score: responders (greater than 75% reduction in PASI from baseline), intermediate-responders (those with greater than 25% and less than 75% reduction in PASI from baseline), and non-responders (less than 25% reduction in PASI from baseline).
Time Frame: 12 Weeks
Measure: Count of Participants; unit: Participants
Groups:
- Etanercept: Patients who received 100 mg Etanercept injections per week for 3 months with recorded PASI score at Week 0 and Week 12 visits.
Arm/Group | Etanercept
Number analyzed (Participants) | 42
Participants
  Responders | 19
  Intermediate Responders | 20
  Non-Responders | 3

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected during the study period time between baseline visit and final visit, 12 weeks.
Description: Adverse events, start date and time, end date, severity, outcome, relation to study drug, relation to study procedure and severity were assessed, collected and recorded in Adverse Event (AE) log by study staff at each visit. The total number of participants at risk includes only those subjects who received study drug at baseline visit. Four subjects consented and withdrew from the study prior to study drug administration; therefore, they were not considered at risk.
Arm/Group | Etanercept
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 1/46
Other Adverse Events (participants affected / at risk) | 9/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept (N=46)
Post-Op Constipation (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept (N=46)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 3 (3)
GI Distress (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-29): https://cdn.clinicaltrials.gov/large-docs/46/NCT01971346/Prot_SAP_000.pdf